CLINICAL TRIAL: NCT06335602
Title: The Evaluation of Traditional Chinese Medicine Intervention for Post-operative Edema After Cruciate Ligament Reconstruction
Brief Title: TCM for Post-operative Edema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YI-WEN HSIEH, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202301283A3
Record Dates: First submitted 2024-03-07; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Acupuncture Treat (Experimental): Low level laser therapy to acupoints related to operation wound, before and after operation
  Interventions: Device: LASER acupuncture
- Laser Acupuncture Sham (Sham Comparator): Low level laser therapy(with Sham device) to acupoints related to operation wound, before and after operation
  Interventions: Device: LASER acupuncture
- Herbal packing (Active Comparator): External application of herbal medicine packing around the operation wound, before and after operation
  Interventions: Device: LASER acupuncture

INTERVENTIONS:
Device: LASER acupuncture — Low level LASER therapy

SUMMARY:
There are loads of research on knee surgery, including surgical methods, rehabilitation strategies, and complication prevention. Whether it is general surgery or endoscopic surgery, there may be postoperative joint swelling, which may last for several weeks depending on the patient's condition. Therefore, reducing swelling as soon as possible is important in post-operative treatment. Swelling of the knee joint may increase soft tissue tension, causing pain and discomfort, and affecting the range of motion and functional recovery of the joint. It may also affect wound healing and increase the risk of complications such as infection and thrombosis. Most clinical research related to traditional Chinese medicine focuses on reducing pain, and little attention is paid to reducing swelling, relatively. Nevertheless most relevant literatures discuss total knee replacement surgery.

Cruciate ligament surgery is very common in sports medicine orthopedics. It is expected that ordinary patients get function recovery quickly after surgery, and athletes can return to play as soon as possible. This study is a prospective study, with partially double-blinded, randomized controlled study design. The investigators are aiming to TCM intervention for knee swelling after cruciate ligament surgery, and evaluation of postoperative swelling and functional improvement. TCM intervention methods are laser acupuncture and external application of herbal medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign informed consent
2. Age between 18-50 years old male and female patients
3. First time receiving cruciate ligament reconstruction
4. Willing to accept TCM intervention and follow up

Exclusion Criteria:

1. Repeat surgical intervention
2. History of serious acupuncture syncope
3. History of severe allergic response of herbal packing or drug-induced dermatitis
4. History of other diseases that cause knee joint swelling, such as rheumatoid arthritis, knee joint infection, gouty arthritis, connective tissue disease, tumor, or cardiac/renal failure.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Leg girth measurement | before operation, day of operation, 1 day/ 2weeks/ 4weeks after operation
  lower limb multiple girth measurement

SECONDARY OUTCOMES:
VAS | before operation, day of operation, 1 day/ 2weeks/ 4weeks after operation
  general scoring of pain
WOMAC | before operation, day of operation, 1 day/ 2weeks/ 4weeks after operation
  specific scoring of joint pain
Tegner score | before operation, day of operation, 1 day/ 2weeks/ 4weeks after operation
  scoring of joint activity